CLINICAL TRIAL: NCT02733939
Title: Åldrande: en Innovativ Och teknologistödd hemmiljö för äldre Patienter Med Alzheimers Sjukdom, TECH@HOME.
Brief Title: Technologies to Reduce Caregiver Burden for Informal Caregivers of People With Dementia
Acronym: TECH@HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-4913
Record Dates: First submitted 2016-03-10; First posted 2016-04-12 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Dementia
Keywords: technology; informal care; caregiver burden
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technology intervention (Experimental): Patients randomized in the intervention group will receive a technical home monitoring kit for 12 months. The kits will be composed of a control unit and a set of sensors that immediately notify caregivers, through their phones, of any potential risks for the person with dementia. The kit will have home leaving sensors, bed occupancy sensors, smoke and water leak sensors, automatic lights, and other interactive functions. These devices will be connected to a single-board microcontroller that will transmit alarm messages to the caregivers in case of need.
  Interventions: Device: Home monitoring kit
- Usual care (No Intervention): Patients receiving usual care, as provided to people with dementia in Southern Sweden can vary. In the target area, people with dementia usually receive comparable pharmaceutical treatment depending on the dementia type, as prescribed by a general practitioner or a specialist at a memory clinic. The social worker from the Municipality ("Biståndshandläggaren") where the person resides, together with the district nurse, have a meaningful role in tailoring the care plan by mediating access to other care services such as respite care homes, home help and (dementia) nurse home visits. Use of such services depends on the specific needs of the person with dementia, which can also be unrelated to dementia, but rather dependent upon concomitant health and social issues.

INTERVENTIONS:
Device: Home monitoring kit — The home monitoring kits notify the caregivers about potentially dangerous situations, such as when the person with dementia:
  * leaves the home without notice, since this might occur in a moment of disorientation;
  * leaves a water tap open;
  * forgets something on the stove;
  * gets out of bed during the night and doesn't come back within a certain time interval;
  * never goes to the bathroom in 24 hours;
  * never opens refrigerator door in 24 hours.
  Depending on the personal choice of the study participants, the kit will also :
  * automatically turn on a light to help avoid a fall during the night;
  * alert the caregiver when the temperature in the house falls or rises excessively;
  * act as burglar alarm in some areas of the home.
  Arms: Technology intervention

SUMMARY:
This randomized controlled trial aims to recruit a total of 320 dyads composed by persons with dementia living in community settings and their primary informal caregivers. In the intervention group, persons with dementia will have a home monitoring kit installed in the household while participants in the control group will receive their usual care. The kit includes home leaving sensors, smoke and water leak sensors, bed sensors as well as automatic lights that monitor the individual's behavior. Alerts (text message and/or phone call) will be sent to the caregiver if anything unusual occurs. All study participants will receive three home visits by project administrators that have received project specific training in order to harmonize data collection. These will take place at enrollment and 3 and 12 months following installation of the home kits. At every home visit, a standardized questionnaire will be administered to all study participants to assess their health, quality of life and resource utilization. The primary outcome of this trial is the amount of informal care support provided by primary informal caregivers to the Person with Dementia.

DETAILED DESCRIPTION:
While the enormous technological progress made in recent years has put technologies, such as mobile devices and smart phones, in the reach of many, innovators in dementia care are just starting to explore the full potential of these developments to transform them into valuable products and services for users. There is indeed a lack of studies that evaluate the effectiveness and cost-effectiveness of these new technologically-enriched interventions targeted at people with dementia. Previous large scale evaluations of the impact of telemedicine and telecare, such as the Whole Demonstrator System in the United Kingdom, did not include people with dementia despite Alzheimer's disease being one of the most burdensome diseases in Europe.

This randomized controlled trial aims to evaluate the effects of new technologies on caregiver burden by reducing the time spent in supervision. The trial builds on previous promising results from the UP-TECH project in Italy (https://clinicaltrials.gov/ct2/show/NCT01700556) . The technologies used in TECH@HOME will include similar, but improved, home monitoring kits potentially leading to a greater impact on caregivers' caring conditions. In addition, while the UP-TECH study did not allow the researchers to estimate the impact of the technology as a "stand-alone" intervention (the monitoring kits were only given in combination with case-management support), TECH@HOME will overcome this limitation thanks to the possibility to compare a group of technology users vs. non-users. Results from this intervention in dementia care in Sweden hold the potential to inform regional and national policy makers in Sweden and beyond.

ELIGIBILITY:
Inclusion Criteria for the person with dementia:

* a diagnose of major neurocognitive disorders with mild to moderate severity (DSM-5) (following the new diagnostic criteria of the American Psychiatric Association;
* A score between 10 and 24 on the Mini-Mental State Examination (MMSE-SR);
* A score between 1 and 5 in the Global Deterioration Scale (GDS)
* Community dwelling;
* Able to speak and understand Swedish;
* Have at least one informal caregiver.

Exclusion Criteria for the person with dementia:

* Lack of informed consent;
* Being fully dependent on caregiver support for the Activities of Daily Living;
* Presence of severe diseases associated with a life expectancy of less than 6 months;
* Intention of moving to institutionalized care during the study period;
* Unwillingness to use technological devices for home assistance and safety;
* Being enrolled in another ongoing trial;
* Substance use disorder (DSM-5).

Specific inclusion criteria for the informal caregiver are:

* Lack of informed consent;
* Unwillingness to use technological devices for home assistance and safety;
* Presence of severe diseases associated with a life expectancy of less than 6 months;
* Being already enrolled in another ongoing trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in time spent in informal care at month 3 | 3 months
  The amount of informal care provided by caregivers to the persons with dementia, considered as a proxy of the caregiver burden, will be measured in hours/week and assessed using a specific section of the Resource Utilization in Dementia (RUD) instrument.
Change from baseline in time spent in informal care at month 12 | 12 months
  The amount of informal care provided by caregivers to the persons with dementia, considered as a proxy of the caregiver burden, will be measured in hours/week and assessed using a specific section of the Resource Utilization in Dementia (RUD) instrument.

SECONDARY OUTCOMES:
Change from baseline in Quality of Life of the person with dementia at month 3 | 3 months
  Quality of life of the person with dementia will be measured using the QOL-AD instrument which has been developed in collaboration with caretakers, caregivers and experts in dementia care to ensure validity. Previous studies suggest that the instrument's validity and reliability are satisfactory in a study population of people with dementia.
Change from baseline in Quality of Life of the person with dementia at month 12 | 12 months
  Quality of life of the person with dementia will be measured using the QOL-AD instrument which has been developed in collaboration with caretakers, caregivers and experts in dementia care to ensure validity. Previous studies suggest that the instrument's validity and reliability are satisfactory in a study population of people with dementia.
Change from baseline in Fear of falling at month 3 | 3 months
  Fear of falling of the person with dementia will be measured using the 16-item Falls Efficacy Scale-International (FES-I). The evaluation of the Swedish version of the instrument showed high internal reliability also among people with cognitive impairment.
Change from baseline in Fear of falling at month 12 | 12 months
  Fear of falling of the person with dementia will be measured using the 16-item Falls Efficacy Scale-International (FES-I). The evaluation of the Swedish version of the instrument showed high internal reliability also among people with cognitive impairment.
Change from baseline in Quality of life of the caregiver at month 3 | 3 months
  Quality of life of the caregiver will be assessed using the EQ-5D-3L. This standardized instrument to measure health outcomes has been used and validated in previous Swedish studies.
Change from baseline in Quality of life of the caregiver at month 12 | 12 months
  Quality of life of the caregiver will be assessed using the EQ-5D-3L. This standardized instrument to measure health outcomes has been used and validated in previous Swedish studies.
Change from baseline in Caregiver anxiety at month 3 | 3 months
  Caregiver anxiety will be assessed using the anxiety component of the Hospital Anxiety and Depression Scale (HADS). HADS is a 14-item scale; seven of the items relate to anxiety and seven relate to depression; each item is a Likert scale rated from 0 to 3, and this means that the overall score for either anxiety or depression will be range from 0 to 21.
Change from baseline in Caregiver anxiety at month 12 | 12 months
  Caregiver anxiety will be assessed using the anxiety component of the Hospital Anxiety and Depression Scale (HADS). HADS is a 14-item scale; seven of the items relate to anxiety and seven relate to depression; each item is a Likert scale rated from 0 to 3, and this means that the overall score for either anxiety or depression will be range from 0 to 21.
Change from baseline in Caregiver burden using the Zarit Burden Inventory (ZBI) at month 3 | 3 months
  The Zarit Burden Inventory (ZBI) will be used to measure the level of caregiver burden. This is the instrument most consistently used in dementia caregiving research, and it is often used to measure the change of caregiver burden over time, resulting from the progression of the disease severity of the care recipient or from interventions aimed at reducing burden. The revised version of the Zarit with 22 items will be used.
Change from baseline in Caregiver burden using the Zarit Burden Inventory (ZBI) at month 12 | 12 months
  The Zarit Burden Inventory (ZBI) will be used to measure the level of caregiver burden. This is the instrument most consistently used in dementia caregiving research, and it is often used to measure the change of caregiver burden over time, resulting from the progression of the disease severity of the care recipient or from interventions aimed at reducing burden. The revised version of the Zarit with 22 items will be used.
Domestic accidents at month 3 | 3 months
  This outcome is measured as the total count of domestic accidents, defined as: 1) accidental falls, 2) cuts, 3) episodes of wandering outside the home, 4) burns and fires in the home, 5) flooding which will be assessed using an ad-hoc form.
Domestic accidents at month 12 | 12 months
  This outcome is measured as the total count of domestic accidents, defined as: 1) accidental falls, 2) cuts, 3) episodes of wandering outside the home, 4) burns and fires in the home, 5) flooding which will be assessed using an ad-hoc form.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Chiatti, PhD, Principal Investigator — Lund University and Italian National Institute on Health and Ageing (INRCA)
Locations (1):
- Memory Clinic, Hospital of Ängelholm, Ängelholm, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malmgren Fange A, Schmidt SM, Nilsson MH, Carlsson G, Liwander A, Dahlgren Bergstrom C, Olivetti P, Johansson P, Chiatti C; TECH@HOME Research Group. The TECH@HOME study, a technological intervention to reduce caregiver burden for informal caregivers of people with dementia: study protocol for a randomized controlled trial. Trials. 2017 Feb 9;18(1):63. doi: 10.1186/s13063-017-1796-8. PMID 28183323